CLINICAL TRIAL: NCT03305354
Title: Mobile Intervention to Improve Functional Health and Community Engagement of Post-9/11 Veterans With Chronic Insomnia: Does Enhancing Physical Activity Help?
Brief Title: Mobile Intervention to Improve Functional Health and Community Engagement of Post-9/11 Veterans With Chronic Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Quigley, Research Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-09-10
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chronic Insomnia
Keywords: mobile health; physical activity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTI app intervention (Experimental): Cognitive Behavioral Therapy for Insomnia delivered for 6 weeks via the CBT-I Coach app with use guided by a self-management guide
  Interventions: Behavioral: CBTI app intervention
- CBTI app+Physical Activity Intervention (Active Comparator): Cognitive Behavioral Therapy for Insomnia delivered for 6 weeks via the CBT-I Coach app with use guided by a self-management guide plus self-management guidance on increased step counts
  Interventions: Behavioral: CBTI app intervention; Behavioral: Physical Activity intervention

INTERVENTIONS:
Behavioral: CBTI app intervention — Self-management guided use of a mobile app called the CBT-I Coach to teach sleep hygiene and enhance sleep
Behavioral: Physical Activity intervention — Self-management guided motivation to increase physical activity by increasing daily step counts
  Arms: CBTI app+Physical Activity Intervention

SUMMARY:
Veterans of the most recent wars in Afghanistan and Iraq (collectively, post 9/11 Veterans) have notable sleep problems including chronic insomnia. Here, the investigators plan to compare two groups of veterans with insomnia: (1) one group that completes a 6 week self-management-guided use of a mobile app based on cognitive behavioral therapy for insomnia (CBTI alone) and (2) one group that completes a 6 week combined self-management-guided use of the mobile CBTI app in addition to a physical activity (PA) intervention (CBTI + PA). The investigators hypothesize that the group receiving the adjunctive 6-week PA intervention will have better subjective and objective sleep, higher step counts, and better functional health and social and community integration than those receiving CBTI alone. This pilot work will provide evidence to guide the design of a future randomized controlled trial.

DETAILED DESCRIPTION:
To determine if the addition of physical activity (PA) to (CBTI) can further enhance sleep, physical activity, functioning, or social engagement over and above self-management use of a CBTI app alone, the investigators will randomly assign post-9/11 veteran participants with chronic, functionally impairing insomnia to either (1) a self-management-based use of an app based on cognitive behavioral therapy for insomnia (CBTI; CBTI alone arm) or to (2) a self-management-based use of the CBTI app + a physical activity (PA) intervention (CBTI + PA) that includes PA monitoring (via a Fitbit device) with individualized goal-setting to encourage increased daily steps across the 6 weeks. For the PA goal, the investigators will attempt to get all participants to at least the typical 10,000 daily steps goal cited as a strong predictor of positive health outcomes (Choi, Pak, & Choi, 2007). The investigators will tailor the step goals based on the person's initial level of daily steps, and increment step goals weekly to maximize motivation and enhance the likelihood that the participant can meet the goal.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals will be US military Veterans
* Eligible veterans will have served in the military during the post-9/11 period
* Eligible veterans will have chronic, functionally impairing insomnia (i.e., at baseline veterans must have an Insomnia Severity Index score > 10 with insomnia duration of at least 1 month, and impaired daytime functioning.
* Eligible individuals must be willing to use devices (e.g., Fitbit, WatchPAT)provided by the study team.
* Eligible individuals may have mild or moderate obstructive sleep apnea (as determined by one out of either of two nights with a WatchPAT-based Apnea-Hypopnea Index [AHI] <= 30 events/hour of sleep).

Exclusion Criteria:

* Periodic leg movements
* Circadian rhythm disorder
* Use of medications or health issues (e.g., permanent pacemaker, sustained non-sinus cardiac arrhythmias, finger deformity, etc.) that would interfere with the use of the WatchPAT sleep monitor
* Severe obstructive sleep apnea (as determined by one out of either of two nights with a WatchPAT-based Apnea-Hypopnea Index [AHI] > 30 events/hour of sleep)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index Total Score | 6 weeks (Immediate post-intervention)
  Total score on the Insomnia Severity Index
Pittsburgh Sleep Quality Index Total Score | 6 weeks (Immediate post-intervention)
  Total score on the Pittsburgh Sleep Quality Index Total Score

SECONDARY OUTCOMES:
Objective Sleep Efficiency | 6 weeks (Immediate post-intervention)
  Time spent in bed divided by time spent asleep as measured by the WatchPAT sleep monitor
Daily step counts | 6 weeks (Immediate post-intervention)
  Daily step counts as measured by a Fitbit device

OTHER OUTCOMES:
Functional Outcomes of Sleep | 6 weeks (Immediate post-intervention)
  Functional Outcomes of Sleep Questionnaire total score (10 item version)
Social Engagement | 6 weeks (Immediate post-intervention)
  Total score on the Lubben Social Network Scale
Community Engagement | 6 weeks (Immediate post-intervention)
  Total score on the Community Integration Questionnaire
Physical Functional Health | 6 weeks (Immediate post-intervention)
  Physical Function score from the Veteran's RAND-12 scale
Mental Functional Health | 6 weeks (Immediate post-intervention)
  Mental Function score from the Veteran's RAND-12 scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Quigley, PhD, Principal Investigator — Northeastern University
Locations (1):
- Edith Nourse Rogers Memorial VA Hospital, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaitz J, Robinson SA, Petrakis BA, Reilly ED, Chamberlin ES, Wiener RS, Quigley KS. Veteran Acceptance of Sleep Health Information Technology: a Mixed-Method Study. J Technol Behav Sci. 2023;8(1):57-68. doi: 10.1007/s41347-022-00287-x. Epub 2022 Dec 13. PMID 36530383
- [Derived] Reilly ED, Robinson SA, Petrakis BA, Gardner MM, Wiener RS, Castaneda-Sceppa C, Quigley KS. Mobile Intervention to Improve Sleep and Functional Health of Veterans With Insomnia: Randomized Controlled Trial. JMIR Form Res. 2021 Dec 9;5(12):e29573. doi: 10.2196/29573. PMID 34889746